CLINICAL TRIAL: NCT04203225
Title: Comparison of 2 Application Techniques for LET (Lidocaine 4%; Epinephrine 0.1%; Tetracaine 0.5%) Gel Used Prior to Simple Laceration Repair in Children
Brief Title: Comparison of Two Application Techniques for LET Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Kelly Young, Senior Physician, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30846-01
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Lacerations; Pain, Procedural; LET
MeSH Terms: conditions — Lacerations; Pain, Procedural | interventions — Epinephrine; Tetracaine; Gels; Linear Energy Transfer

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized study; patients are randomized to one of two groups
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Investigator and nurse applied intervention and masked the intervention from the care provider. Separate nurse not caring for the patient, blinded to the intervention, brought in to obtain pain score (outcome)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single LET (Active Comparator): One (single) application of LET topical gel [Lidocaine (4%), Epinephrine (0.1%), and Tetracaine (0.5%)] applied for 30 minutes
  Interventions: Drug: LET Lidocaine (4%), Epinephrine (0.1%), and Tetracaine (0.5%) topical gel
- Triple LET (Experimental): Three applications of LET topical gel, one applied every 10 minutes
  Interventions: Drug: LET Lidocaine (4%), Epinephrine (0.1%), and Tetracaine (0.5%) topical gel

INTERVENTIONS:
Drug: LET Lidocaine (4%), Epinephrine (0.1%), and Tetracaine (0.5%) topical gel — Topical anesthetic
  Other Names: LET

SUMMARY:
Comparison of anesthetic efficacy of Lidocaine (4%), Epinephrine (0.1%), and Tetracaine (0.5%) topical gel (LET) applied three times for 10 minutes each time vs. once for 30 minutes prior to suturing simple lacerations in children aged 7-17 years.

DETAILED DESCRIPTION:
Randomized single-blinded clinical trial with convenience sampling of the anesthetic efficacy of a single 30-minute application vs three 10-minute applications of Lidocaine (4%), Epinephrine (0.1%), and Tetracaine (0.5%) topical gel (LET) prior to suturing simple lacerations in children aged 7-17 years seen in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* Simple <= 3cm lacerations requiring suturing (as decided by clinician care providers)
* Plan to suture with simple interrupted sutures

Exclusion Criteria:

* Lacerations involving the hands, feet, genitals, tongue, mucus membranes, nose, ears, or occurring over joints
* Patients whose primary language was neither English nor Spanish
* Developmentally delayed or disabled patient such that they were unable to give a pain score
* Patients requiring procedural sedation or anxiolysis with oral or intranasal midazolam

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly D Young, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital of Orange County, Orange, California
  - Harbor-UCLA Medical Center, Torrance, California

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Derived] Siembieda J, Heyming T, Padlipsky P, Young KD. Triple Versus Single Application of Lidocaine, Epinephrine, and Tetracaine for Laceration Repair in Children. Pediatr Emerg Care. 2022 Feb 1;38(2):e472-e474. doi: 10.1097/PEC.0000000000002631. PMID 35100752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Convenience sample, pediatric emergency departments at Harbor-UCLA Medical Center and Children's Hospital of Orange County
Period: Overall Study
Arm/Group | Single LET | Triple LET
Started | 21 | 27
Completed | 21 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single LET | Triple LET | Total
Number analyzed (Participants) | 21 | 27 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 27 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (3.1) | 10.3 (2.6) | 10.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 16 | 23 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 14 | 22 | 36
  Race/Ethnicity: White | 2 | 2 | 4
  Race/Ethnicity: Black | 1 | 1 | 2
  Race/Ethnicity: Asian / Pacific Islander | 1 | 1 | 2
  Race/Ethnicity: Other | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 21 | 27 | 48
Laceration location [Count of Participants; unit: Participants]
  Face/Scalp | 18 | 20 | 38
  Arm | 0 | 2 | 2
  Leg | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Score
Description: Pain score self-rated by patient on 100m Visual Analog Pain scale, minimum value 0, maximum value 100, higher scores equal more pain (worse outcome)
Time Frame: Immediately on placement or attempt at placement of first suture
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Single LET | Triple LET
Number analyzed (Participants) | 21 | 27
mm | 16 (17) | 16 (24)

2. Secondary Outcome: Need for Additional Local Anesthetic
Description: Need for additional infiltrated local anesthetic (lidocaine)
Time Frame: At any time during suturing procedure, time frame is duration of procedure, generally 10-20 minutes, less than one hour. Determined by chart review immediately after procedure completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Single LET | Triple LET
Number analyzed (Participants) | 21 | 27
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: During the patient's emergency department visit until time of discharge.
Arm/Group | Single LET | Triple LET
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/27
Other Adverse Events (participants affected / at risk) | 0/21 | 0/27

LIMITATIONS AND CAVEATS:
* Unable to blind the patient and nurse caring for the patient
* Wide age range from which we recruited patients
* We included children only age 7 years and older in order to be able to obtain a self-reported VAS pain score
* Majority of lacerations were on the face / scalp
* Sustaining a laceration and then being in an emergency department is already traumatic for young children; could interfere with pain scores

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT04203225/Prot_SAP_000.pdf